CLINICAL TRIAL: NCT01232322
Title: Pulmicort Respules 0.25/0.5 Specific Clinical Experience Investigation for Long-term Use in Pediatrics
Brief Title: Pulmicort Respules 0.25/0.5 Specific Clinical Experience Investigation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5257L00014
Record Dates: First submitted 2010-10-31; First posted 2010-11-02 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Bronchial Asthma
Keywords: bronchial asthma; Pulmicort Respules; long term use; pediatrics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmicort Respules: Those with an exposure

SUMMARY:
The purpose of this study is to investigate the safety and efficacy for long term treatment of the drug in children aged 6 months and < 5 years on bronchial asthma in daily clinical usage.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Pulmicort Respules for the first time due to bronchial asthma
* Children of >= 6 months and < 5 years old age at the start of study treatment

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients treated with Pulmicort respules for the first time due to bronchial asthma and children of >=6months and <5 years old age at the start of study treatment
Sampling Method: Non-Probability Sample
Enrollment: 633 (Actual)
Dates: Start 2006-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Range of 3 years
Effects on growth rate | Range of 3 years
  Variation of the height/weight from the baseline.
Effects on the adrenal cortical function. | Range of 3 years
  Symptoms of adrenal cortical function suppression before and after the treatment with Pulmicort.
Effects on development of infections. | Range of 3 years
  Existence and type of infections.

SECONDARY OUTCOMES:
Clinical course under Pulmicort long-term use
  Validation of the frequency of asthmatic attack, level of the asthmatic attack, daily life, night sleep from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yoshida Shigeru, MD, Study Director — AstraZeneca